CLINICAL TRIAL: NCT03389724
Title: Prevention of Chemotherapy Induced Cardiotoxicity in Children With Bone Tumors and Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCHE -AML0001
Record Dates: First submitted 2017-12-13; First posted 2018-01-04 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Cardiotoxicity; Acute Myeloid Leukemia in Children; Bone Tumor
MeSH Terms: conditions — Cardiotoxicity; Bone Neoplasms | interventions — Captopril

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized study where all patients presenting to the CCHE with de novo diagnosis of Bone tumor (ES and OS) and AML will be randomized to receive (Intervention arm) or not to receive (Control arm) prophylactic ACE-I with the start of chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group capoten (Intervention arm) (Experimental): Patients will receive prophylactic ACE-I(Capoten®) at day 1 of initiation of chemotherapy and is to be continued for 1 year after the end of treatment. Patients will remain on this arm until they experience any of the study primary or secondary end-point where they will be off-study and will receive cardiotoxicity treatment independently.
  Interventions: Drug: Capoten®
- Group standard treatment (Control arm) (No Intervention): Patients will not receive ACE-I as prophylaxis, and will be monitored and evaluated for first signs of cardiotoxicity based on the above mentioned end-points.

INTERVENTIONS:
Drug: Capoten® — ACE-I (Capoten®) will be given to patients in the Intervention arm with the start of chemotherapy, twice daily at a dose of 0.5 mg/kg/day (divided over 2 doses)
  Other Names: Captopril
  Arms: Group capoten (Intervention arm)

SUMMARY:
Prevention and early detection of chemotherapy-induced cardiotoxicity in children with bone tumors and Acute Myeloid Leukemia by giving capoten

DETAILED DESCRIPTION:
background and rationale: Developing countries bear the greatest burden of childhood cancers as over 90% of the world's children live in these countries. More effective treatment protocols have markedly improved the outcome of childhood cancers. The 5-year overall survival for children with cancer in general has improved from about 30% in 1960s to about 80% currently. Most of current treatment protocols for childhood cancer utilize anthracyclines as an essential chemotherapeutic agent. However, the use of anthracyclines has been limited by their dose dependent cardiotoxic side-effects during and after treatment. Many survivors of anthracycline treatment have long-term problems because of myocardial damage such as impaired left ventricular contractility and cardiomyopathy, which may lead to overt heart failure and an increased risk of death.Anthracycline-induced clinical heart failure (A-CHF) is a major public health concern within the exposed population as it may not be manifested for many years and remains a lifelong threat. It is a particular problem in children treated for cancer because it is hoped that they will survive for several decades after treatment. As survival rates continue to improve, the resources needed to predict, monitor and care for survivors will also continue to increase Several risk factors have been already identified for anthracyclines induced cardiotoxicity. Among the non modifiable risk factors are age at treatment, length of survival, sex, and few genetic factors Other important risk factors include cumulative dose of anthracyclines, rate of administration, concomitant irradiation and chemotherapeutic agents Several approaches have been tried to prevent or minimize cardiotoxicity in cancer patients. Structural modifications of anthracyclines, including liposomal anthracyclines and anthracycline analogs, have been developed with the intention to minimize cardiovascular toxicity. Epirubicin and idarubicin, analogs of doxorubicin and daunorubicin, respectively, are commonly used to treat few types of cancer. The use of liposomal anthracyclines considerably reduces anthracycline cardiotoxicity but does not eliminate it. A recent meta-analysis of two studies found that the rates for both clinical and subclinical heart failure were significantly lower with liposomal anthracyclines than with conventional anthracyclines and that tumor response and overall survival rates did not differ significantly. Both studies were limited in scope because only adult women with metastatic breast cancer were included. No randomized controlled trials comparing liposomal with conventional anthracyclines in children have been published.

Observational studies have shown that prolonged infusion of anthracyclines reduces cardiotoxicity than bolus infusions. However, a randomized controlled trial reported no statistically significant differences in echocardiographic parameters up to 8 years after treatment of patients receiving either continuous infusion or bolus administration.

Dexrazoxane (the only agent proven to reduce acute cardiotoxicity in adults receiving anthracyclines) is not currently recommended in children due to raised concerns of increased incidence of secondary neoplasms.Angiotensin-Converting Enzyme Inhibitors (ACEIs) have shown marked reduction of toxic myocarditis in mouse models ( and have also shown marked decrease in adverse myocardial histopathological changes in mice treated with anthracyclines . Administration of ACEIs as a cardioprotective agent was studied in high risk cancer patients (defined by increased troponin I value) and proven to be effective . The role of ACEIs in prevention of anthracyclines induced cardiotoxicity was not examined before in a randomized controlled setting.

Proper evaluation and early prediction of cardiotoxicity necessitates a consensus on sensitive and specific monitoring methods in the pediatric population. However, several studies have addressed the rapidly evolving issue of cardiotoxicity assessment. Several cardiac biomarkers have been used to monitor and predict cardiotoxicity. Among those markers are: Cardiac Troponin T (cTnT), Cardiac Troponin I (cTnI), Atrial Natriuretic Peptide (ANP), Brain Natriuretic Peptide (BNP), N-terminal pro-BNP (NT-pro-BNP), Serum Lipid Peroxide, and Serum Carnitine. Several systematic reviews have highlighted the difficulty of assessing those biomarkers due to several limitations in performed studies and high variability. Further research is needed to establish the effectiveness of cardiac markers in children, and their link to anthracycline dose, and their use in predicting individual risk for the development and progression of cardiotoxicity .

However, more recent studies have shown that troponins are preferred due to their high sensitivity and specificity, especially when coupled with imaging modalities.

Imaging modalities for diagnosis and follow up of cardiotoxicity are the main gold standard. Echocardiogram (Doppler) is the most commonly used method due its high availability and non invasiveness. Radionuclide Angiocardiography (RNA) including MUGA have also been used. Although RNA studies exhibit lower intra-individual and intra-observer variation when obtaining and analyzing results, but only limited information regarding diastolic function is obtained. RNA's also expose patients to radiation .

A recent study has demonstrated that the use of Tissue Doppler-derived myocardial performance index is a more robust parameter in the detection of ventricular dysfunction caused by doxorubicin when compared to Doppler.

In summary, anthracyclines induced cardiotoxicity continues to be one of the most challenging problems facing children with cancer during and after treatment. No current consensus exists about the best method for early detection and monitoring of cardiotoxicity in children with cancers. Troponins, echocardiography, and tissue Doppler have shown promising results as effective modalities but they need to be further studied especially in this specific population. Several protective agents have also been tried to prevent cardiotoxicity. ACE-Inhibitors have shown promising results in adult cancer patients, but they have not been studied before in the pediatric population.

Objectives of the Study:

Aim of the Study: (Instructions: state the goal you need to achieve) Prevention and early detection of chemotherapy-induced cardiotoxicity in children with bone tumors and Acute Myeloid Leukemia.

Specific Objectives: (Instructions: state the details of each objective that will finally lead to achievement of the goal)

1. To determine the incidence of early and late (subclinical and clinical) cardiotoxicity during anthracycline chemotherapy in children with Bone tumors & AML, and associated risk factors.
2. To determine the role of ACE-I in preventing chemotherapy-related cardiotoxicity
3. To determine the role of troponin I (TnI) as an early marker of cardiac toxicity .
4. To measure the accuracy of other radiological techniques for early detection of cardiotoxicity like Tissue Doppler Imaging (TDI) and Speckle-tracking Echo (STE).

Secondary Objectives: (Instructions: these are subsidiary objectives that could be studied during the course of the project but are not the main objectives of the study, they are optional and vary according to the type of the study).

1. To standardize the monitoring, evaluation and grading of cardiotoxicity based on CTCAE,v4 and Modified Ross Classification.
2. To standardize Reporting of cardiac functions using electronic sheets on Cerner for documentation.

ELIGIBILITY:
Inclusion Criteria:

* All Acute Myeloid Leukemia and Bone Tumors patients (Osteosarcoma and Ewing's Sarcoma) who didn't receive chemotherapy will be included in the study.
* Written Informed Consent from parents/guardian

Exclusion Criteria:

* Patients who received chemotherapy before starting of the study
* Patients with history of cardiac impairment, (existing or congenital heart disease).
* Patients who show intolerance or contra-indications to ACE-I.
* Patients developing acute (< 2 weeks) cardiotoxicity after the first high-dose chemotherapy (HDC) course.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 245 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
To determine the effect of ACE-I in preventing chemotherapy-related cardiotoxicity using both investigation techniques: Troponin I level and cardiac imaging ( TTE, TDI, STE). | 3 years
  ALL patients will be subjected to the following cardiac imaging ( TTE, TDI, STE) at the each time intervals of the study.
  Plasma troponin I (TnI) concentration will be measured for all the patients at the each time intervals of the study.
To determine the role of Troponin I (TnI) as an early marker of cardiac toxicity | 3 years
  Troponin I (TnI) concentration is to be determined by a fluorometric enzyme immunoassay analyzer (Stratus CS, Dade Behring, Miami, Fla) with a functional sensitivity of 0.03 g/L; the cutoff level was 0.08 ng/mL.
  Plasma troponin I (TnI) concentration will be measured in both groupsas follows :
  * Early TnI: TnI concentration will be measured before and soon after each cycle of HDC. Determination of early TnI consists of a curve of assays (2ml blood sample): baseline initially, before & after immediately, and 12 and 24 hours after the end of Anthracycline chemotherapy infusion.This sequence will be repeated with each cycle of therapy containing Anthracycline. For each patient, the highest TnI value will be considered for each chemotherapy cycle.
  * Late TnI: TnI value also is to be determined at the end of treatment and 2, 3, 6, and 12 months after end of treatment in both groups.
To measure the accuracy of other radiological techniques for early detection of cardiotoxicity like Tissue Doppler Imaging (TDI) and Speckle-tracking Echo (STE). | 3 years
  Patients will be evaluated Clinically for cardiac functions using ECG , conventional echo, Tissue Doppler Imaging (TDI) and SpeckelTracking Echocardiography STE , before each chemotherapy cycle maximum one week given

CONTACTS AND LOCATIONS:
Overall Officials: Zeniab salah, MD, Principal Investigator — Children's Cancer Hospital Egypt 57357 Cairo, Egypt
Locations (1):
- Children's Cancer Hospital Egypt 57357 Cairo, Egypt, Cairo, Egypt